CLINICAL TRIAL: NCT04083391
Title: Is Hamstring Flexibility Affected in Chronic Ankle Instability
Brief Title: Flexibility Deficit in Chronic Ankle Instability
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abd Elhady Samy Abu Mandour, Principal investigator, Cairo University
Other Study IDs: P.T.REC/012/001312
Record Dates: First submitted 2019-08-23; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Chronic Ankle Instability
Keywords: chronic ankle instability; Hamstring; flexibility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — 21 patients with CAI and 21 participants without ankle sprain injury
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CAI group: assessment had been done to this group that include patients with ankle sprain injury from more than one year and complain with repetitive injuries, giving way and instability feelings
- non injured ankle group: assessment had been done to this group that include control participants had not injured their ankle before and matched with CAI in age, gender, dominant side

SUMMARY:
chronic ankle instability could be associated with some proximal deficits as in hip and knee regions. these deficits include alternations in motor neurons pools excitability, muscle strength, kinematics and kinetics. this study add muscle inflexibility to the preciouse literature.

DETAILED DESCRIPTION:
Background: influence of a localized injury in a distal joint on the function of proximal muscles is an important consideration in assessment and treatment of musculoskeletal injuries. Up to the investigator's knowledge, there is no study assess flexibility changes in CAI. Objectives: The objective of this study is to investigate Hamstring flexibility in CAI. Material and methods: The study conducted on 42 subjects with unilateral CAI and controls had measure of hamstring flexibility using digital inclinometer during passive knee extension test .Results: Revealed statistical and clinical significant difference between non-injured control group and CAI group with decreased hamstring flexibility in the later. Conclusion: CAI subjects have proximal muscular affection include hamstring tightness which may alter sacroiliac joint stability and subsequently back pain.

ELIGIBILITY:
Inclusion Criteria:

* The control group was self-reported to be healthy
* Had no ankle injury history
* Matched with CAI patients in gender, dominance side and simulated injured side
* CAI group had a self-report of a past history of unilateral ankle inversion injury since at least more than 1 year before the study onset which required a period of protected weight bearing and/or immobilization at least one day
* Patient reported a tendency for the ankle to give way and/or recurrent ankle sprain
* Perceives that the ankle was chronically weaker, more painful and/or less functional than the other ankle or than before first

Exclusion Criteria:

* Had a history of lower extremity injury
* Surgery or fracture
* History of low back dysfunction that required medical or surgical intervention within the last year, Current participation in formal or informal rehabilitation
* History of hamstring strain
* Bilateral ankle sprain injury
* Ankle injury within 3 months of participation
* History of ankle fracture and any neuromuscluskeletal disease could affect the condition.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Outpatients clinic faculty of physical therapy Cairo university
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2016-05-07 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
Hamstring muscle flexibility | throughout the study average 1 year
  angle between tibia and femur during passive knee extension test

CONTACTS AND LOCATIONS:
Overall Officials: Afaf Tahoon, Master, Study Chair — assistant lecturer faculty of physical therapy Cairo university

IPD SHARING:
Plan to Share IPD: No
IPD had been planed to be shared with research team only through specific username and password

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT04083391/Prot_SAP_000.pdf